CLINICAL TRIAL: NCT06505928
Title: A Parallel-group, Randomized, Open-label Clinical Trial of Hepalatide for Injection in Patients With Chronic Hepatitis D.
Brief Title: A Clinical Trial of Hepalatide for Injection in Patients With Chronic Hepatitis D
Acronym: L47-HD-MN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L47-HD-MN
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis D
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Intervention Model Description: This is a three-arm, parallel-group, randomized, open-label, delayed-controlled phase IIb clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hepalatide 2.1mg (Experimental): hepalatide 2.1mg/d, s.c. for 48 weeks
  Interventions: Drug: hepalatide
- Hepalatide 4.2mg (Experimental): hepalatide 4.2mg/d, s.c. for 48 weeks
  Interventions: Drug: hepalatide
- delayed treatment groups (No Intervention): delayed treatment for 48 weeks

INTERVENTIONS:
Drug: hepalatide — hepalatide of 2.1 mg/d or 4.2mg/d s.c. treatment for 48 weeks
  Other Names: L47
  Arms: Hepalatide 2.1mg; Hepalatide 4.2mg

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of L47 in the treatment of chronic hepatitis D. Patients with compensated CHD who satisfy the eligibility criteria are stratified by the presence or absence of liver cirrhosis and randomized into three groups at a 1:1:1 ratio. The subjects will receive continuous L47 (2.1 mg/d and 4.2 mg/d, s.c.) treatment for 48 weeks (groups A and B), or delayed treatment for 48 weeks (group C). Primary endpoint evaluation will be performed after the subjects complete the 48-week treatment.

DETAILED DESCRIPTION:
This is a three-arm, parallel-group, randomized, open-label, delayed-controlled phase IIb clinical trial. The study flow chart is shown in Fig. 1.2.1. CHD patients with compensated liver function who satisfy the eligibility criteria are stratified by the presence or absence of liver cirrhosis and randomized into the 2.1 mg group, 4.2 mg group, and delayed treatment group at a 1:1:1 ratio (Table 1.1). The subjects will receive continuous L47 (2.1 mg/d and 4.2 mg/d, s.c.) treatment for 48 weeks (groups A and B), or delayed treatment for 48 weeks (group C). The 1st interim analysis will be performed when all subjects complete the Week12 visit to determine the optimal dose for the extended treatment period following the trial. The 2nd interim analysis will be performed when all subjects complete the Week24 visit. Upon completion of the 48th week of treatment, the primary endpoint was assessed, and the trial was officially concluded.

After the conclusion of the trial, all subjects in each group entered the extension treatment period and were all treated continuously with the L47 optimal dose for 96 weeks. After the extension treatment ended, all groups discontinued the medication and were observed for 48 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subjects aged 18-65 years (both inclusive);
* 2. Subjects with positive HBsAg and/or HBV DNA for at least 6 months ("CHB");
* 3. Subjects with positive serum anti-HDV antibody before or at screening or with positive HDV RNA for at least 6 months before screening ("CHD");
* 4. Subjects with positive and quantifiable HDV RNA before enrollment;
* 5. 1 × ULN < ALT < 10 × ULN;
* 6. Subjects who should be treated with nucleoside/nucleotide reverse transcriptase inhibitors at enrollment or after enrollment according to the guidelines for the treatment of hepatitis D (compensated cirrhosis with detectable HBV DNA, or HBV DNA > 2000 IU/mL in patients without cirrhosis) and consent to the use of entecavir for the treatment of chronic hepatitis B;
* 7. Subjects who do not plan a pregnancy within 3 years (women who are not pregnant or lactating, and males who agree to take effective contraceptive measures throughout the treatment period and for 3 months after the last dose);
* 8. Subjects exhibiting good compliance to the study protocol;
* 9. Subjects who understand the ICF and agree to sign it.

Exclusion Criteria:

* 1. Subjects suffering from severe decompensated liver fibrosis or decompensated liver cirrhosis with a Child-Pugh score > 7;
* 2. Decompensated liver disease: Direct bilirubin > 1.2 x ULN or prothrombin time > 1.2 x ULN or serum albumin < 35 g/L;
* 3. Abnormal hematology findings: White blood cell count (WBC) < 3 × 109/L, neutrophil count < 1.5 × 109/L or platelet count < 60 × 109/L;
* 4. Creatinine clearance < 60 mL/min;
* 5. Subjects who have any of the following conditions:

  1. History of current or past decompensated liver diseases (including coagulopathy, hepatic encephalopathy, and variceal bleeding);
  2. Comorbidity of underlying diseases such as severe infection, heart failure and chronic obstructive pulmonary disease, and other severe diseases;
  3. Diabetes mellitus and hypertension not effectively controlled (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg);
  4. Current or previous uncontrolled epilepsy or psychiatric disorders;
  5. History of solid organ transplantation;
  6. Evidence of active or suspected malignancies or history of malignancies, or untreated premalignant lesions within the past 5 years (except for successfully treated cervical carcinoma in situ at least 1 year before screening, and successfully treated basal cell carcinoma and squamous cell carcinoma [≤ 3 cases of resected skin cancer within 5 years before screening ]), or history of liver cancer;
  7. History of alcohol abuse or drug addiction at present or within 6 months prior to participation in this study; 6. Subjects co-infected with hepatitis A, C, or E virus or with uncontrolled HIV co-infection (those with positive HCV antibody but negative HCV RNA at screening are eligible for enrollment. HIV-infected patients may be enrolled if cluster of differentiation 4 (CD4) cell count is > 500/mL and HIV RNA is below the limit of detection for at least 12 months);
* 7. Presence of one or more other known primary or secondary liver diseases, such as alcoholism, autoimmune hepatitis, malignancies involving the liver, hemochromatosis, other congenital or metabolic diseases affecting the liver, congestive heart failure, or other serious cardiopulmonary diseases, excluding hepatitis B;
* 8. Subjects with one or more autoimmune diseases, immune-related extrahepatic manifestations (such as vasculitis, purpura, arteritis nodosa, peripheral neuropathy, and glomerulonephritis), or a history of requiring regular use of systemic corticosteroids (inhaled corticosteroids are allowed) or other immunosuppressive agents;
* 9. Subjects who have used interferon within 6 months before screening;
* 10. Subjects who have used L47 or Bulevirtide within 3 months;
* 11. Allergy to entecavir;
* 12. Pregnant or breastfeeding women;
* 13. Subjects who participated in other drug clinical trials within 30 days before randomization;
* 14. Subjects who are receiving prohibited treatment at screening that cannot be discontinued;
* 15. Subjects who cannot comply with the study protocol and complete all procedures as scheduled, or have significant abnormalities in other laboratory or auxiliary examinations, which render them ineligible for this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
compound response | Week 48
  Decrease in HDV RNV by ≥ 2 log10 from baseline and ALT normalization

SECONDARY OUTCOMES:
HDV RNA below LLOQ | Week 48
  The incidence of subjects with HDV RNA lower than LLOQ.
Decrease in HDV RNA by ≥ 2 log10 from baseline or undetectable HDV RNA | Week 48
  The incidence of subjects with Decrease in HDV RNA by ≥ 2 log10 from baseline or undetectable HDV RNA
Decrease in HDV RNA from baseline | Week 48
  HDV RNA reduction from baseline.
ALT normalization | Week 48
  The rate of ALT relapse in subjects.
Decrease in ALT from baseline | Week 48
  ALT reduction from baseline.
Changes in subjects' METAVIR system scores from baseline. | Week 48
  The METAVIR score is a test used to determine the degree of inflammation and necrosis in the liver biopsy, as well as the extent of fibrosis. The degree of liver fibrosis is divided into five grades from F 0 to F4. The degree of inflammatory activity in liver tissue is divided into four grades from A0 to A3. Higher score means worse outcome.
  When the liver tissue inflammation and necrosis score decreased by ≥2 points compared with baseline (the change of inflammatory activity A value compared with baseline was ≤ -2 points), and there was no increase in liver fibrosis score; Or the liver fibrosis score decreased by ≥1 point (fibrosis stage F value change from baseline ≤ 0 points)，it means Liver tissue response.
Change in fibrosis 4 (FIB-4) index from baseline | Week 48
  Fibrosis 4（FIB-4）Index is a non-invasive method for assessing liver fibrosis in patients with chronic liver disease. The FIB-4 index is <1.45, indicating no significant liver fibrosis or only 2nd degree or lower liver fibrosis. And the FIB-4 index>3.25 indicates that the degree of liver fibrosis is 3-4 or higher.
Change in Child-Pugh score from baseline | Week 48
  Child-Pugh scores is a test that determines the scope and severity of liver failure as well as the prognosis for the patient. Three categories "A, B and C " indicate the severity of liver breakdown on the Child-Pugh rating scale. The higher the scale, the more serious outcomes.
Change in Model for End-Stage Liver Disease (MELD) score from baseline | Week 48
  R = 9.6 \* ln(serum creatinine in mg/dl) + 3.8 \* ln(bilirubin in mg/dl) + 11.2 \* ln(INR) + 6.4 \* cause (cause: cholestasis and alcoholic cirrhosis = 0, viral and other causes of cirrhosis = 1). The higher the R value, the greater the risk, and the lower the survival rate.
The incidence rate of Liver-related endpoint events. | Week 240
  The incidence of Liver-related endpoint events such as cirrhosis, hepatic decompensation, HCC, liver transplantation, liver-related death.

CONTACTS AND LOCATIONS:
Overall Officials: Oyunbileg Janchiv, Principal Investigator — National Cacer Center of Monglia
Locations (2):
- Mongolia (2):
  - National cancer canter of Monglia, Ulaanbaatar
  - National Center for Communicable Diseases, Ulaanbaatar